CLINICAL TRIAL: NCT05715463
Title: Achieving Equity in Inflammatory Arthritis Care: An Adaptive Trial To Understand and Address Social Determinants of Health
Brief Title: Rheumatology-based Adaptive Intervention for Social Determinants and Health Equity
Acronym: RAISE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Candace Hillary Feldman, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022P003268
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis; Palindromic Arthritis; Juvenile Rheumatoid Arthritis; Ankylosing Spondylitis; Sacroiliitis; Psoriatic Arthritis; Mixed Connective Tissue Disease; Lupus; Enteropathic Arthropathies; Systemic Sclerosis; Sjogren's Syndrome; Sicca Syndrome; Inflammatory Arthritis; Undifferentiated Connective Tissue Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Juvenile; Spondylitis, Ankylosing; Sacroiliitis; Arthritis, Psoriatic; Mixed Connective Tissue Disease; Scleroderma, Systemic; Sjogren's Syndrome; Arthritis; Undifferentiated Connective Tissue Diseases

STUDY DESIGN:
Intervention Model Description: This will be an adaptive intervention. After six months, Individuals who do not respond to Arm 1, as measured by no improvement in SDoH-related needs and/or an outpatient no show or same day cancellation, will increase to the Arm 2 intervention for the next 6 months (see Schema). Patients in Arm 1 who do respond will graduate and then complete a follow-up set of questionnaires at 12 months. Patients in Arm 2 or Arm 3 who adequately respond and have had their SDoH-related needs addressed will graduate and receive a follow-up set of questionnaires at 12 months. Individuals in Arm 2 who continue to have one or more no show and/or continue to have SDoH-related needs will be ramped up to Arm 3. Individuals in Arm 3 with the same scenario will remain in Arm 3 for another 6 months. Data will be collected for 12 months (at baseline, 6 and 12 months) for participants in all arms including those who graduate at 6 months, to determine if the response was sustained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Other): Arm 1 is the control arm which will receive the standard of care resource sheets.
  Interventions: Other: Resource sheets
- Arm 2 (Experimental): Arm 2 will receive the assistance of a community resource specialist (CRS)- an individual without formal medical training with community-based expertise.
  Interventions: Other: Community Resource Specialist
- Arm 3 (Experimental): Arm 3 will receive the assistance of a bilingual (English and Spanish) nurse patient navigator with nursing training and additional rheumatology-specific training.
  Interventions: Other: Nurse Navigator

INTERVENTIONS:
Other: Resource sheets — Arm 1 is the control arm which will receive the standard of care resource sheets. Patients in this arm will receive cultivated resource sheets for any SDoH-related needs that they screen positive for or request additional information on.
  Arms: Arm 1
Other: Community Resource Specialist — The CRS will help guide patients to the necessary community-based resources to help address their specific SDoH needs that impact their health and their ability to access sustained, high quality medical care. This may include forms to arrange for subsidized transportation to and from medical appointments or applications for Section 8 housing. The community resource specialist will reach out to patients in Arm 2 a minimum of 2 times per month, with more interactions guided by patients needs. All outreach attempts and contacts will be documented in EPIC and in REDCap. Actions taken by the CRS will be shared with members of the patient's healthcare team as appropriate (with EPIC notes routed to the rheumatologist and primary care provider, and if indicated and relevant, a social worker, nutritionist, prior CRS, nurse or mental health provider if previously involved in the patient's care).
  Arms: Arm 2
Other: Nurse Navigator — The nurse navigator will both work with the CRS to connect the patient with community-based resources, independently connect the patient with relevant resources, and also help coordinate the patient's medical care and mental health needs. The nurse patient navigator will conduct her own needs assessment (the nurse navigator high risk assessment questionnaire at the time of the first conversation with the patient, originally developed as part of the MGB integrated care management program) and her actions will be guided by their responses. She will reach out to patients a minimum of 2 times per month with an increase in communication around patient appointments as reminders, and more frequent communication on a case-by-case basis depending on active illnesses, frequency of outpatient appointments, and needs of the patient. All outreach attempts and contact will be documented in EPIC and in REDCap and similar to the CRS, be shared via EPIC with the care team as indicated.
  Arms: Arm 3

SUMMARY:
Social determinants of health (SDoH), defined by the World Health Organization as "the conditions in which people are born, grow, work, live and age and the wider set of forces and systems shaping the conditions of daily life" are estimated to be responsible for nearly 90 percent of a person's health outcomes. SDoH are key contributors to racial, ethnic and socioeconomic disparities in care healthcare access and health outcomes. The goal of this clinical trial is to identify patients with inflammatory arthritis or with a systemic rheumatic condition with arthritis who may respond to the simplest and least expensive intervention to address their SDoH-related needs- a tailored list of resources, those who benefit from a community-based resource specialist to help address specific needs, and those who require a nurse-trained navigator to help both coordinate the services provided by the community-based specialist, and their medical and mental health care and needs. The main questions the clinical trial aims to answer are:

1. To test the efficacy of a rheumatology clinic-based nurse navigator and community resource specialist to reduce appointment no-shows and same-day cancellations in patients with systemic rheumatic conditions with arthritis.
2. To examine the cost-effectiveness of each of the different study interventions for individuals with systemic rheumatic conditions with arthritis with SDoH-related needs using questionnaires and cost-related care metrics.

Participants will be randomly assigned to 1 of 3 arms. In Arm 1, patients will receive a cultivated list of resources related to the needs that patients indicate on the social determinants of health questionnaire. Arm 1 is the control arm which receives the current standard of care. In Arm 2, patients will receive the assistance of a community resource specialist (CRS) - an individual without formal medical training with community-based expertise. In Arm 3, patients will receive the assistance of a nurse patient navigator with additional systemic rheumatic condition-specific training who will work with the CRS.

After 6 months, patients who do not respond to Arm 1 will move to Arm 2. Patients who do not respond to Arm 2, will move to Arm 3. Patients who do not respond to Arm 3 will remain in Arm 3. Patients who respond to any arm will graduate the program at 6 months. The patients who do not respond be in their new arm for 6 months. At 12 months, all patients remaining in the study will graduate.

DETAILED DESCRIPTION:
Social determinants of health (SDoH), defined by the World Health Organization as "the conditions in which people are born, grow, work, live and age and the wider set of forces and systems shaping the conditions of daily life" are estimated to be responsible for nearly 90 percent of a person's health outcomes. SDoH are key contributors to racial, ethnic and socioeconomic disparities in care healthcare access and health outcomes. Among patients with chronic rheumatic conditions, SDoH including poverty, insurance status, and inadequate access to care have been shown to contribute to delayed diagnoses, frequent emergency department visits, medication nonadherence, worse quality of life, increased disease-related damage and poorer outcomes. Individuals with inflammatory arthritis often require complex, costly medication regimens and suffer from a high burden of comorbid conditions and physical disabilities. They face unique healthcare challenges including a high risk of care fragmentation from multiple subspecialty providers and medications that are both expensive and challenging to adhere to as prescribed. The role of SDoH on the care and outcomes of patients with inflammatory arthritis is understudied but living conditions, socioeconomic status and neighborhood income have been shown to contribute to treatments received and the likelihood of remission at 12 months. Disparities in inflammatory arthritis care and outcomes are likely multifactorial and involve both delayed access to subspecialty care as well as ongoing barriers to sustained, high quality care once referred. Separate comprehensive interventions are required to address the challenges at every stage of care.

Our ongoing quality improvement initiative aims to collect and document social determinants of health data for people with inflammatory arthritis across this multi-hospital system. In this initiative the investigators developed a standard of care where patients have their needs assessed and if they indicate that they would like information to help address these needs, they are sent resource lists. A community resource specialist is also available when indicated to help address needs. In this study, the investigators aim to test different interventions to address the needs that the investigators uncover using the SDoH screening protocol. Using an adaptive strategy, patients with SDoH-related needs and appointment no shows in the past, will be randomized to one of three arms, with the ability to change arms if they do not improve in their assigned arm. Cost-effectiveness analyses will also be conducted.

Using an adaptive intervention, this trial will help identify patients who may respond to the simplest and least expensive intervention - a tailored list of resources, those who benefit from a community-based resource specialist to help address specific SDoH-related needs, and those who require a nurse-trained navigator to help both coordinate the services provided by the community-based specialist, and their medical and mental health care and needs. A cost effectiveness analysis of the interventions will be conducted. The knowledge gained by this trial will help guide care and advocacy for vulnerable populations both in resource poor settings and at major medical centers that have not previously allocated the services needed to care for the highest risk populations. The overall goal of this study is to provide these essential data to advocate for a scalable, sustainable program to meet the needs of the most vulnerable patients with chronic rheumatic conditions with arthritis that can be scaled to other chronic systemic rheumatic diseases and other complex, subspecialty-managed conditions.

Specific Aims:

1. To conduct a randomized controlled trial with an adaptive intervention to test the efficacy of a rheumatology clinic-based nurse patient navigator and community resource specialist intervention to reduce appointment no shows. This intervention will allow for an understanding of these needs and test three strategies to begin to address them. The investigators anticipate that all of the interventions will benefit to some degree through connection to resources. The investigators currently have no data as to whether one type of intervention is better than another for patients with systemic rheumatic conditions with arthritis and therefore, the investigators are testing two types of navigator interventions with the ultimate goal of determining the most beneficial and cost-effective intervention for high-risk patients based on their specific needs. The adaptive nature of the intervention will allow the study team to study this further and will allow for as many individuals as possible to derive potential benefit from this study.
2. To examine the cost-effectiveness of each of the different study arms for individuals with systemic rheumatic conditions with arthritis with SDoH-related needs using the ED-5D questionnaire and cost-related care metrics.

Subjects will be identified using the EHR (EPIC review, EDW, RPDR), and through BRASS. Rheumatologists will also be asked to refer patients who they feel may be appropriate. Patients will be recruited via patient gateway, by mail or by rheumatologist referral. Rheumatologists and the clinic nursing team will also be given fact sheets and recruitment letters that they can give to patients they feel might be interested in participating. If a letter is sent to a patient via gateway, via mail, or introduced by the rheumatologist, if the patient does not opt out, at least one week later, a member of the study team will call the patient to follow up. If they cannot be reached by phone but have a rheumatology clinic visit >=1 week after the letter is sent, a member of the research team may approach them in clinic to see if they might be interested in learning more about the study. The research assistants will be responsible for identifying and recruiting individuals beginning at the date of IRB approval. Communication for recruitment will occur in-person, through secure messaging in the EHR, through secure email (unless the patient opts out of secure email) and via the telephone. The patients enrolled in this study may have frequent appointment no shows and some may more frequently come to the Emergency Department or be admitted (either at BWH or at Faulkner). Therefore, the research team may approach patients for consent while they are in the ED or on an inpatient floor if unable to reach them by phone or in clinic. Similarly, the community resource specialist or nurse navigator may interact with the patients when they are in the ED or admitted due to the nature of their role (especially for those patients with frequent acute care use, who may also be those with the greatest SDoH-related needs).

Prior studies have demonstrated that individuals who experience poverty and increased SDoH-related needs have an increased burden of rheumatic conditions, more severe outcomes, and increased care fragmentation. As such, the investigators aim to enroll individuals in this intervention who are at highest risk for adverse outcomes and high acute care use to address SDoH-related needs and improve receipt of outpatient care. The study team aims to include a racially and ethnically diverse patient population in this study. The investigators expect that more females than males will be enrolled because rheumatic conditions are more prevalent among females. The investigators expect that the majority of patients enrolled will be English-speaking given the ethnicity distribution of patients served in the rheumatology clinics at BWH (<10% identify as Latinx). To allow for the inclusion of Spanish-speaking patients, however, the study team has included translated materials.

The investigators anticipate recruiting 258 patients with systemic rheumatic conditions with arthritis across Mass General, Brigham and Faulkner hospitals and satellite rheumatology clinics to participate in the intervention components of this trial (N=86 per arm). Patients will be associated with the study in Epic so the study staff is notified if patients go to the ED or are hospitalized. The primary analysis will be intention-to-treat, and since the primary outcome metric can be obtained from the EHR, even if patients are lost to follow-up, the study team will still be able to collect these data. However, given the vulnerability of the patient population and potential loss to follow-up, the investigators will have statistical power to detect a clinically meaningful difference in medication and appointment adherence between the two intervention arms with 156 total patients (N=52 per arm) using a per protocol design, and examining secondary outcomes that require survey completion.

Study Team Interactions with Subjects Patients who agree to participate will be randomized to one of three arms. Arm 1 is the control arm which will receive the standard of care resource sheets. Patients in this arm will receive cultivated resource sheets for any SDoH-related needs that they screen positive for or request additional information on. Arm 2 will receive the assistance of a community resource specialist (CRS)- an individual without formal medical training with community-based expertise, who will help guide patients to the necessary community-based resources to help address their specific SDoH needs that impact their health and their ability to access sustained, high quality medical care. This may include forms to arrange for subsidized transportation to and from medical appointments or applications for Section 8 housing. The community resource specialist will reach out to patients in Arm 2 a minimum of 2 times per month, with more interactions guided by patients' needs. All outreach attempts and contacts will be documented in EPIC and in REDCap. Arm 3 will receive the assistance of a bilingual (English and Spanish) nurse patient navigator with nursing training and additional rheumatology-specific training who will both work with the CRS to connect the patient with community-based resources, independently connect the patient with relevant resources, and also help coordinate the patient's medical care and mental health needs. The nurse patient navigator will conduct her own needs assessment (the nurse navigator high risk assessment questionnaire at the time of the first conversation with the patient, originally developed as part of the MGB integrated care management program) and her actions will be guided by their responses. She will reach out to patients a minimum of 2 times per month with an increase in communication around patient appointments as reminders, and more frequent communication on a case-by-case basis depending on active illnesses, frequency of outpatient appointments, and needs of the patient. All outreach attempts and contact will be documented in Epic and REDCap and shared via EPIC with the care team as indicated.

Reassignments after 6 months After six months, individuals who do not respond to Arm 1 will be reassigned to the Arm 2 intervention (CRS). Response will be determined by >=1 appointment no shows or same day cancellations during the 6-month period and/or persistence of >=1 SDoH-related need that has not been addressed. Individuals without any no shows who had their needs addressed will graduate and will receive follow-up surveys at 12 months. Patients in Arm 2 or Arm 3 with no appointment now shows and who have had their SDoH-related needs addressed will graduate and complete follow-up surveys at 12 months. If individuals in Arm 2 had >=1 no show and/or persistent SDoH-related needs, they will be reassigned to Arm 3 (nurse navigator). If individuals in Arm 3 had >=1 no show and/or persistent SDoH-related needs, they will remain in Arm 3 for another 6 months. All individuals will complete 12-month surveys.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking
* 18+ years of age
* diagnosis of a systemic rheumatic condition with arthritis
* 1+ prior no-show(s) or same day cancellation(s) to an ambulatory care provider in the past year
* 1+ social determinants of health needs on Mass General Brigham questionnaire (excluding unemployment and education)
* Receiving rheumatology care at a Mass General Hospital, Brigham and Women's Hospital or Faulkner Hospital affiliated clinic

Exclusion Criteria:

* Incarcerated individuals
* Indicated through our EHR that they do not want to be contacted for research
* Patients already actively enrolled in an integrated care management program through their primary care provider
* Medical complexity that requires urgent nursing involvement and thus not medically appropriate for randomization

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient no-shows | -12 months through +12 months
  Patient no-shows will be measured through EPIC data from EDW, manual chart review and RPDR. The outcome will measure number of times that a patient has been designated 'no show' to an appointment with an ambulatory care provider.

SECONDARY OUTCOMES:
Reduction of Social Determinants of Health-related needs in institution-created questionnaire | -12 months through +12 months
  Patient social determinants of health-related needs will be measured through the institution-created social determinants of health questionnaire. The social determinants of health questionnaire has 11 questions for patient to indicate if they do or do not have certain needs. The patient can respond yes or no to having a lack of transportation to and from appointments. The patient is given a scale of never true, sometimes true and often true for 2 questions regarding food insecurity, The patient can indicate that they do or do not have housing today (or choose not to answer), and they can indicate how many times they moved in the last year as 0, 1, or 2+. For the remaining questions regarding housing, paying for utilities, paying for medications, unemployment, education and child or family care, the patient can respond yes, no or choose not to answer. Responses of yes indicate the patient has a need, and no indicates that they do not have a need.
Reduction of Social Determinants of Health-related needs in EHR data | -12 months through +12 months
  Patient social determinants of health-related needs will be measured through patient EHR data.
Medication adherence through patient questionnaire | 0 through +12 months
  Patient medication adherence will be measured through the patient self-completed questionnaire. The patient indicates how many days they missed a dose of their medication between 1 and 30. The following question asks how often patients took their medications as they were supposed to and can indicate between never and always. The final questions asks how well the patient took their medications as they were supposed and they can respond between very poor to excellent.
Medication adherence through medication refill data | 0 through +12 months
  Patient medication adherence will be measured through patient refill data from Epic.
Acute care use overall | 0 through +12 months
  Patient acute care use for overall will be measured through EHR data for emergency department visits and hospitalizations.
Acute care use for avoidable conditions | 0 through +12 months
  Patient acute care use for overall will be measured through EHR data for emergency department visits and hospitalizations.
Treat-to-target metrics | 0 through +12 months
  Patient treat-to-target measures will be measured through patient-reported disease activity metrics, specifically the Routine Assessment of Patient Index Data 3 (RAPID3) which includes pain, global assessment of health and physical function. The scores range from 0 to 10.0 with 0 -1.0 defined as near remission, 1.3 - 2.0 as low severity, 2.3 - 4.0 as moderate severity and 4.3 - 10.0 as high severity.
Patient trust in providers | 0 through + 12 months
  Patient trust will be measured through patient trust questionnaire. The scale is scored 5 - 1 with strongly agree, agree, neutral, disagree and strongly disagree. The higher the patient score, the higher the trust in the provider.
Self efficacy | 0 through +12 months
  Patient self efficacy will be measured through a self efficacy questionnaire. For 6 questions the patient can respond between 0 and 10 with 0 indicating not confident at all and 10 being totally confident. The final score is the mean of the items on the survey. Higher numbers indicate higher self efficacy and lower numbers indicate lower self efficacy.
Patient anxiety & depression | 0 through +12 months
  Patient anxiety and depression will be measured through the Patient Health Questionnaire 4 (PHQ4). Items 1 and 2 address patient anxiety and items 3 and 4 address patient depression. Both anxiety and depression score on a scale of 1 - 6, with a scale of 3 or more on either scale being a positive screen.
Patient stress | 0 through +12 months
  Patient stress will be measured through the perceived stress scale 4 (PSS-4). The individual questions are measure 0 - 4, with the lowest score being 0 and the highest score being 16. Higher scores are correlated with higher stress.
Disability metric | 0 through +12 months
  Patient disability and health will be measured through EuroQol 5D (EQ5D) questionnaire. The first 5 questions are measured 1 to 5 with the higher number corresponding to a higher level of disability. The final question is on a scale of 0 to 100 with lower scores corresponding to worse health.
Patient discrimination | 0 through +12 months
  Patient discrimination will be measured through Everyday Discrimination questionnaire. The patient will indicate which areas of discrimination they have experienced. The more items that are checked, the greater discrimination they have experienced.
Patient satisfaction | 0 through +12 months
  Patient satisfaction will be measured through Patient Satisfaction questionnaire 18 (PSQ 18). Each question is measured on a scale of 1 to 5, with 1 being strongly agree and 5 being strongly disagree. After question-specific scoring, the higher the overall score should reflect higher patient satisfaction.
Inflammatory Arthritis Checklist | 0 through +12 months
  Patient preventative measures will be tracked through the inflammatory arthritis checklist.
Lupus Checklist | 0 through +12 months
  Patient preventative measures will be tracked through the inflammatory arthritis checklist.
Literacy | 12 months
  Patient literacy will be assessed by asking how comfortable patients feel in completing medical forms by themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Candace H Feldman, MD, MPH, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States